CLINICAL TRIAL: NCT04154956
Title: Randomized, Open-label, Phase 3 Study of SAR408701 Versus Docetaxel in Previously Treated, Metastatic Nonsquamous, Non-small-cell Lung Cancer Patients With CEACAM5-positive Tumors
Brief Title: SAR408701 Versus Docetaxel in Previously Treated, Carcinoembryonic Antigen-related Cell Adhesion Molecule 5 (CEACAM5) Positive Metastatic Non-squamous Non-small-cell Lung Cancer Patients
Acronym: CARMEN-LC03
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC15858; U1111-1233-0781 (Registry Identifier: ICTRP); 2024-515101-26-00 (Registry Identifier: CTIS); 2019-001273-81 (EudraCT Number)
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Results first posted 2024-11-01 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Non-small Cell Lung Cancer Metastatic
MeSH Terms: interventions — tusamitamab ravtansine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SAR408701 (tusamitamab ravtansine) (Experimental): Participants received tusamitamab ravtansine 100 milligrams per square meter (mg/m^2) by intravenous (IV) infusion, once every 2 weeks (Q2W) until objective progressive disease (PD), unacceptable adverse event/toxicity, upon participant's request to stop treatment, or Investigator decision, whichever occurred first (maximum exposure: 147 weeks).
  Interventions: Drug: SAR408701
- Docetaxel (Active Comparator): Participants received docetaxel 75 mg/m^2 by IV infusion, once every 3 weeks (Q3W) until objective PD, unacceptable adverse event/toxicity, upon participant's request to stop treatment, or Investigator decision, whichever occurred first (maximum exposure: 115 weeks).
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: SAR408701 — Pharmaceutical form: Concentrate for solution for intravenous infusion Route of administration: intravenous (IV) infusion
  Arms: SAR408701 (tusamitamab ravtansine)
Drug: Docetaxel — Pharmaceutical form: Concentrate for solution for intravenous infusion Route of administration: IV infusion
  Other Names: TAXOTERE
  Arms: Docetaxel

SUMMARY:
Primary Objectives:

* Study was designed with multiple primary endpoints analyzed on randomized participants at the time of the cut-off date for each given analysis (progression free survival [PFS] and overall survival [OS])
* Study success was defined either on PFS or OS
* The primary objective was to determine whether tusamitamab ravtansine improves the progression free survival (PFS) when compared to docetaxel in participants with metastatic non-squamous non-small-cell lung cancer (NSCLC) expressing CEACAM5 greater than or equal to 2+ in intensity in at least 50% of the tumor cell population and previously treated with standard-of-care platinum-based chemotherapy and an immune checkpoint inhibitor (ICI)
* The primary objective was to determine whether tusamitamab ravtansine improves the overall survival (OS) when compared with docetaxel in participants with metastatic non-squamous NSCLC expressing CEACAM5 greater than or equal to 2+ in intensity in at least 50% of the tumor cell population and previously treated with standard-of-care platinum-based chemotherapy and an immune checkpoint inhibitor.

Secondary Objectives:

* Compared the objective response rate (ORR) of tusamitamab ravtansine with docetaxel
* Compared the health-related quality of life (HRQOL) of tusamitamab ravtansine with docetaxel
* Evaluated the safety of tusamitamab ravtansine compared to docetaxel
* Assessed the duration of response (DOR) of tusamitamab ravtansine as compared with docetaxel

DETAILED DESCRIPTION:
The median expected duration of study per participant was estimated as median 9 months in docetaxel arm (1 month for screening, 4 months for treatment, and 4 months for the EOT and follow-up visits) and 12.5 months in SAR408701 arm (1 month for screening, 6.5 months for treatment, and 5 months for end of treatment follow-up).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age or above (or country's legal age of maturity if above 18 years) and signed the informed consent.
* Histologically or cytologically proven diagnosis of non-squamous NSCLC with metastatic disease at study entry; progression after platinum-based chemotherapy and immune checkpoint inhibitor.
* Participants with carcinoembryonic antigen-related cell adhesion molecule (CEACAM) 5 expression of greater than or equal to 2+ in archival tumor sample (or if not available, fresh biopsy sample) involving at least 50% of the tumor cell population as demonstrated prospectively by central laboratory via immune histochemistry (IHC).
* At least one measurable lesion by RECIST v1.1 as determined by local site investigator /radiologist assessment.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* A female participant who agreed to use highly effective contraceptive methods during and for at least 7 months after the last dose of study intervention.
* A male participant who agreed to use highly effective contraception methods during and for at least 6 months after the last dose of study intervention.

Exclusion Criteria:

* Participants with untreated brain metastases and history of leptomeningeal disease. if previously treated brain metastases no documentation of non-progressive disease in brain by imaging performed at least 4 weeks after CNS directed treatment and at least 2 weeks prior to the first dose of study intervention.
* Significant concomitant illnesses, including all severe medical conditions that would impair the participation in the study or interpretation of the results.
* History within the last 3 years of an invasive malignancy other than the one treated in this study, with the exception of resected/ablated basal or squamous-cell carcinoma of the skin or carcinoma in situ of the cervix, or other local tumors considered cured by local treatment.
* Non-resolution of any prior treatment related toxicity to less than grade 2 according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version (V) 5.0, except for alopecia, vitiligo and active thyroiditis controlled with hormonal replacement therapy
* History of known acquired immunodeficiency syndrome (AIDS) related illnesses or known HIV disease requiring antiretroviral treatment, or unresolved viral hepatitis
* Previous history of and/or unresolved corneal disorders. The use of contact lenses was not permitted.
* Concurrent treatment with any other anticancer therapy.
* Prior treatment with docetaxel or maytansinoid derivatives (DM1 or DM4 antibody drug conjugate) or any drug targeting CEACAM5.
* Contraindicated the use of corticosteroid premedication.
* Previous enrollment in this study and current participation in any other clinical study involving an investigational study treatment or any other type of medical research.
* Poor bone marrow, liver or kidney functions
* Hypersensitivity to any of the study interventions, or components thereof (EDTA), or drug (paclitaxel, polysorbate 80) or other allergy that, in the opinion of the Investigator, contraindicated participation in the study.

The above information was not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2026-03-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (169):
- United States (8):
  - Florida Cancer Specialists South Division- Site Number : 8400020, Fort Myers, Florida
  - Florida Cancer Specialists North Division- Site Number : 8400019, St. Petersburg, Florida
  - Ca & Hem Center Of W Michigan- Site Number : 8400016, Grand Rapids, Michigan
  - Roswell Park Cancer Institute Site Number : 8400011, Buffalo, New York
  - Lankenau Hospital Cancer Center- Site Number : 8400017, Wynnewood, Pennsylvania
  - Renovatio Clinical- Site Number : 8400032, El Paso, Texas
  - Renovatio Clinical - Site Number : 8400013, The Woodlands, Texas
  - Medical College of Wisconsin- Site Number : 8400006, Milwaukee, Wisconsin
- Argentina (7):
  - Investigational Site Number : 0320009, CABA, Buenos Aires
  - Investigational Site Number : 0320012, Capital Federal, Buenos Aires
  - Investigational Site Number : 0320003, Viedma, Río Negro Province
  - Investigational Site Number : 0320001, Buenos Aires
  - Investigational Site Number : 0320004, Buenos Aires
  - Investigational Site Number : 0320014, Córdoba
  - Investigational Site Number : 0320002, Salta
- Australia (3):
  - Investigational Site Number : 0360002, Blacktown, New South Wales
  - Investigational Site Number : 0360003, Waratah, New South Wales
  - Investigational Site Number : 0360001, Woolloongabba, Queensland
- Belgium (6):
  - Investigational Site Number : 0560006, Anderlecht
  - Investigational Site Number : 0560004, Edegem
  - Investigational Site Number : 0560005, Ghent
  - Investigational Site Number : 0560001, Leuven
  - Investigational Site Number : 0560003, Liège
  - Investigational Site Number : 0560002, Woluwe-Saint-Lambert
- Brazil (6):
  - Centro Regional Integrado De Oncologia - CRIO- Site Number : 0760002, Fortaleza, Ceará
  - ~Instituto De Oncologia Parana- Site Number : 0760008, Curitiba, Paraná
  - Centro Avancado de Oncologia CECAN - Liga Contra o Cancer- Site Number : 0760026, Natal, Rio Grande do Norte
  - Clínica de Oncologia Reichow Site Number : 0760023, Blumenau, Santa Catarina
  - Hospital de Base Sao Jose do Rio Preto Site Number : 0760001, São José do Rio Preto, São Paulo
  - Hospital Sirio Libanes- Site Number : 0760018, São Paulo, São Paulo
- Bulgaria (6):
  - Investigational Site Number : 1000008, Burgas
  - Investigational Site Number : 1000010, Pleven
  - Investigational Site Number : 1000007, Plovdiv
  - Investigational Site Number : 1000004, Sofia
  - Investigational Site Number : 1000003, Sofia
  - Investigational Site Number : 1000001, Sofia
- Canada (2):
  - Investigational Site Number : 1240003, Greenfield Park, Quebec
  - Investigational Site Number : 1240010, Montreal, Quebec
- Chile (5):
  - Investigational Site Number : 1520007, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520006, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520009, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Viña del Mar, Región de Valparaíso
- China (29):
  - Investigational Site Number : 1560026, Beijing
  - Investigational Site Number : 1560009, Changchun
  - Investigational Site Number : 1560010, Changchun
  - Investigational Site Number : 1560015, Changsha
  - Investigational Site Number : 1560039, Changsha
  - Investigational Site Number : 1560032, Chengdu
  - Investigational Site Number : 1560038, Chengdu
  - Investigational Site Number : 1560044, Chongqing
  - Investigational Site Number : 1560043, Chongqing
  - Investigational Site Number : 1560024, Fuzhou
  - Investigational Site Number : 1560001, Guangzhou
  - Investigational Site Number : 1560036, Guangzhou
  - Investigational Site Number : 1560037, Guangzhou
  - Investigational Site Number : 1560017, Guangzhou
  - Investigational Site Number : 1560025, Hangzhou
  - Investigational Site Number : 1560033, Hangzhou
  - Investigational Site Number : 1560021, Hangzhou
  - Investigational Site Number : 1560011, Hangzhou
  - Investigational Site Number : 1560005, Harbin
  - Investigational Site Number : 1560050, Huizhou
  - Investigational Site Number : 1560047, Jinan
  - Investigational Site Number : 1560023, Nanjing
  - Investigational Site Number : 1560019, Nanjing
  - Investigational Site Number : 1560012, Nanning
  - Investigational Site Number : 1560045, Tianjin
  - Investigational Site Number : 1560006, Wuhan
  - Investigational Site Number : 1560016, Zhanjiang
  - Investigational Site Number : 1560041, Zhengzhou
  - Investigational Site Number : 1560040, Zhengzhou
- France (13):
  - Investigational Site Number : 2500010, Bordeaux
  - Investigational Site Number : 2500008, Caen
  - Investigational Site Number : 2500006, Créteil
  - Investigational Site Number : 2500007, Grenoble
  - Investigational Site Number : 2500001, Marseille
  - Investigational Site Number : 2500013, Montpellier
  - Investigational Site Number : 2500011, Paris
  - Investigational Site Number : 2500014, Paris
  - Investigational Site Number : 2500009, Pierre-Bénite
  - Investigational Site Number : 2500003, Rennes
  - Investigational Site Number : 2500012, Saint-Herblain
  - Investigational Site Number : 2500002, Saint-Mandé
  - Investigational Site Number : 2500004, Villejuif
- Germany (2):
  - Investigational Site Number : 2760002, Essen
  - Investigational Site Number : 2760001, Heidelberg
- Greece (5):
  - Investigational Site Number : 3000005, Athens
  - Investigational Site Number : 3000001, Athens
  - Investigational Site Number : 3000003, Heraklion
  - Investigational Site Number : 3000004, Ioannina
  - Investigational Site Number : 3000006, Thessaloniki
- Hungary (3):
  - Investigational Site Number : 3480003, Budapest
  - Investigational Site Number : 3480007, Budapest
  - Investigational Site Number : 3480005, Kaposvár
- Israel (3):
  - Investigational Site Number : 3760001, Haifa
  - Investigational Site Number : 3760002, Kfar Saba
  - Investigational Site Number : 3760003, Petah Tikva
- Italy (5):
  - Investigational Site Number : 3800004, Ravenna, Emilia-Romagna
  - Investigational Site Number : 3800005, Rozzano, Milano
  - Investigational Site Number : 3800003, Orbassano, Torino
  - Investigational Site Number : 3800006, Catania
  - Investigational Site Number : 3800001, Milan
- Japan (17):
  - Investigational Site Number : 3920002, Nagoya, Aichi-ken
  - Investigational Site Number : 3920015, Nagoya, Aichi-ken
  - Investigational Site Number : 3920012, Fukuoka, Fukuoka
  - Investigational Site Number : 3920008, Kurume-shi, Fukuoka
  - Investigational Site Number : 3920016, Sapporo, Hokkaido
  - Investigational Site Number : 3920017, Himeji-shi, Hyōgo
  - Investigational Site Number : 3920006, Kanazawa, Ishikawa-ken
  - Investigational Site Number : 3920005, Yokohama, Kanagawa
  - Investigational Site Number : 3920009, Natori-shi, Miyagi
  - Investigational Site Number : 3920001, Hirakata-shi, Osaka
  - Investigational Site Number : 3920003, Osaka, Osaka
  - Investigational Site Number : 3920013, Osaka Sayama-shi, Osaka
  - Investigational Site Number : 3920004, Sunto-gun, Shizuoka
  - Investigational Site Number : 3920011, Bunkyo-ku, Tokyo
  - Investigational Site Number : 3920018, Mitaka-shi, Tokyo
  - Investigational Site Number : 3920007, Wakayama, Wakayama
  - Investigational Site Number : 3920010, Ube-shi, Yamaguchi
- Investigational Site Number : 4840003, Cuauhtémoc, Mexico City, Mexico
- Netherlands (3):
  - Investigational Site Number : 5280003, 's-Hertogenbosch
  - Investigational Site Number : 5280004, Breda
  - Investigational Site Number : 5280005, Utrecht
- Poland (2):
  - Investigational Site Number : 6160004, Olsztyn, Warmian-Masurian Voivodeship
  - Investigational Site Number : 6160001, Warsaw
- Portugal (5):
  - Investigational Site Number : 6200002, Almada
  - Investigational Site Number : 6200001, Lisbon
  - Investigational Site Number : 6200004, Lisbon
  - Investigational Site Number : 6200005, Porto
  - Investigational Site Number : 6200006, Porto
- Romania (7):
  - Investigational Site Number : 6420008, Alba Iulia
  - Investigational Site Number : 6420009, Brasov
  - Investigational Site Number : 6420003, Bucaresti
  - Investigational Site Number : 6420010, Cluj-Napoca
  - Investigational Site Number : 6420011, Cluj-Napoca
  - Investigational Site Number : 6420012, Otopeni
  - Investigational Site Number : 6420005, Timișoara
- Russia (2):
  - Investigational Site Number : 6430001, Moscow
  - Investigational Site Number : 6430003, Saint Petersburg
- Singapore (2):
  - Investigational Site Number : 7020001, Singapore
  - Investigational Site Number : 7020002, Singapore
- South Korea (7):
  - Investigational Site Number : 4100008, Busan, Busan
  - Investigational Site Number : 4100005, Cheongju-si, North Chungcheong
  - Investigational Site Number : 4100006, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100007, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100003, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100004, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100001, Seoul
- Spain (9):
  - Investigational Site Number : 7240007, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240005, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240001, L'Hospitalet de Llobregat, Barcelona [Barcelona]
  - Investigational Site Number : 7240009, Madrid / Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240006, Pamplona, Navarre
  - Investigational Site Number : 7240002, Madrid
  - Investigational Site Number : 7240004, Málaga
  - Investigational Site Number : 7240011, Seville
  - Investigational Site Number : 7240008, Valencia
- Turkey (Türkiye) (11):
  - Investigational Site Number : 7920008, Adana
  - Investigational Site Number : 7920012, Adana
  - Investigational Site Number : 7920002, Adana
  - Investigational Site Number : 7920011, Ankara
  - Investigational Site Number : 7920005, Istanbul
  - Investigational Site Number : 7920001, Istanbul
  - Investigational Site Number : 7920006, Istanbul
  - Investigational Site Number : 7920007, Izmir
  - Investigational Site Number : 7920010, Izmir
  - Investigational Site Number : 7920014, Kocaeli
  - Investigational Site Number : 7920009, Malatya

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 161 centers in 25 countries from 06 February 2020 to 22 September 2023 (primary completion date). Results are reported as per the primary completion date of 22 September 2023.
Pre-assignment Details: A total of 490 participants were screened, of which 389 participants were randomized in a ratio of 1:1 to either tusamitamab ravtansine or docetaxel arm. The randomization was stratified by Eastern Cooperative Oncology Group (ECOG) performance status (0 versus 1), previous immune checkpoint inhibitor treatment (sequential versus combination with chemotherapy) and geographical region (Asia versus Western Europe + Australia + North America versus Rest of the World [RoW]).
Groups:
- Tusamitamab Ravtansine: Participants received tusamitamab ravtansine 100 milligrams per square meter (mg/m^2) by intravenous (IV) infusion, once every 2 weeks (Q2W) until objective progressive disease (PD), unacceptable adverse event/toxicity, upon participant's request to stop treatment, or Investigator decision, whichever occurred first (maximum exposure: 147 weeks).
Period: Overall Study
Arm/Group | Tusamitamab Ravtansine | Docetaxel
Started | 194 | 195
Randomized and Treated | 194 | 177
Completed | 48 | 52
Not Completed | 146 | 143
Not completed — Death | 109 | 110
Not completed — Not related to Coronavirus disease 2019 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 7
Not completed — Ongoing study treatment at the time of primary analysis | 36 | 25

BASELINE CHARACTERISTICS:
Population: Randomized participants consisted of all participants with a signed main study informed consent form who had a treatment kit number allocated and recorded in the interactive response technology (IRT) database, regardless of whether the treatment kit was used or not.
Groups:
- Tusamitamab Ravtansine: Participants received tusamitamab ravtansine 100 mg/m^2 by IV infusion, once Q2W until objective PD, unacceptable adverse event/toxicity, upon participant's request to stop treatment, or Investigator decision, whichever occurred first (maximum exposure: 147 weeks).
- Docetaxel: Participants received docetaxel 75 mg/m^2 by IV infusion, once Q3W until objective PD, unacceptable adverse event/toxicity, upon participant's request to stop treatment, or Investigator decision, whichever occurred first (maximum exposure: 115 weeks).
- Total: Total of all reporting groups
Arm/Group | Tusamitamab Ravtansine | Docetaxel | Total
Number analyzed (Participants) | 194 | 195 | 389
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (9.2) | 62.3 (9.8) | 62.8 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 86 | 157
  Male | 123 | 109 | 232
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 54 | 58 | 112
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  White | 115 | 94 | 209
  Not reported | 22 | 36 | 58
  Unknown | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from the date of randomization to the date of the first documentation of objective PD as assessed by radiological review committee (IRC) according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) definitions or death due to any cause before the study cut-off date, whichever occurred first. PD was defined as unequivocal progression of existing non-target lesions; appearance of 1 or more new lesions; at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeters (mm).
Time Frame: Tumor assessments performed at screening, and every 8 weeks +/-5 days thereafter, up to 189 weeks
Population: The intent-to-treat (ITT) population consisted of all participants who had given their informed consent and who had a treatment kit number allocated and recorded in the IRT database.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tusamitamab Ravtansine | Docetaxel
Number analyzed (Participants) | 194 | 195
months | 5.39 [3.713 to 6.998] | 5.85 [5.520 to 7.359]
Statistical Analysis 1: Comparison: Tusamitamab Ravtansine vs Docetaxel; Test type: Superiority; p = 0.8204, Log Rank — One-sided significance level was 0.01; Hazard Ratio (HR) = 1.143, 95% CI 2-sided [0.864 to 1.512] — Hazard ratio and confidence intervals (CIs) were computed from a stratified Cox model according to stratification factors as per IRT

2. Primary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from date of randomization to date of death due to any cause.
Time Frame: From date of first study treatment administration (Day 1) until the date of death due to any cause, up to 189 weeks
Population: The ITT population consisted of all participants who had given their informed consent and who had a treatment kit number allocated and recorded in the IRT database.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tusamitamab Ravtansine | Docetaxel
Number analyzed (Participants) | 194 | 195
months | 12.81 [11.795 to 14.160] | 11.53 [8.936 to 15.244]
Statistical Analysis 1: Comparison: Tusamitamab Ravtansine vs Docetaxel; Test type: Superiority; p = 0.1120, Log Rank — One-sided significance level was 0.00174; Hazard Ratio (HR) = 0.846, 95% CI 2-sided [0.644 to 1.109] — Hazard ratio and CIs were computed from a stratified Cox model according to stratification factors as per IRT

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants who had a complete response (CR) or partial response (PR), as best overall response derived from overall response (OR) determined by the IRC per RECIST 1.1. CR was defined as disappearance of all target and non-target lesions, and normalization of tumor marker level. Any pathological lymph nodes (whether target or non-target) must have had reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Tumor assessments performed at screening, and every 8 weeks +/-5 days thereafter, up to 189 weeks
Population: The ITT population consisted of all participants who had given their informed consent and who had a treatment kit number allocated and recorded in the IRT database. Only participants with randomization date ≥8 weeks prior to analysis cut-off date or with early PD prior to the cut-off date are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tusamitamab Ravtansine | Docetaxel
Number analyzed (Participants) | 189 | 187
percentage of participants | 21.7 [16.04 to 28.26] | 24.1 [18.13 to 30.84]
Statistical Analysis 1: Comparison: Tusamitamab Ravtansine vs Docetaxel; Test type: Superiority; p = 0.6972, Cochran-Mantel-Haenszel — P-value is provided for information only, there is no statistical inference based on this P-value; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.55 to 1.42] — Odds ratio and its 2-sided CI were provided from a Cochran-Mantel-Haenszel (CMH) test stratified according to the stratification factors

4. Secondary Outcome: Time to Deterioration (TTD) in Disease-related Symptoms as Determined by European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire and Lung Cancer-specific Module With 13 Items (EORTC QLQ LC-13)
Description: The TTD was defined as the time from baseline (Cycle 1, Day 1) until the first ≥10-point change from baseline up to the end of treatment assessment before the initiation of further anticancer therapy and the analysis cut-off date. For the TTD in disease-related symptoms (cough, dyspnea, pain) from EORTC QLQ LC-13, a deterioration was defined as an increase from baseline score of at least 10 points in any 1 of these 3 symptoms. The EORTC QLQ-LC13 (LC13) is the lung cancer module of the EORTC QLQ-C30 that assesses lung-cancer-associated symptoms (cough, dyspnea, pain, hemoptysis) and side-effects from conventional chemotherapy and radiotherapy (sore mouth, hair loss, dysphagia and neuropathy). The EORTC QLQ-LC13 contains 13 items. Items on the LC13 were scored using the LC13 scoring algorithms which standardize the raw scores to a 0-100 range. Lower scores indicate lower symptomology/symptom burden (lower scores better).
Time Frame: Predose on Day 1 of Cycle 1, then on Day 1 of every 2 docetaxel Cycles, or every 3 tusamitamab ravtansine Cycles (i.e., every 6 weeks) up to 30 days after the last dose of study drug administration, up to 151 weeks
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tusamitamab Ravtansine | Docetaxel
Number analyzed (Participants) | 194 | 195
months | 2.83 [2.103 to 4.304] | 1.87 [1.544 to 2.793]
Statistical Analysis 1: Comparison: Tusamitamab Ravtansine vs Docetaxel; Test type: Superiority; p = 0.0157, Log Rank — P-value is provided for information only, there is no statistical inference based on this P-value; Hazard Ratio (HR) = 0.729, 95% CI 2-sided [0.546 to 0.972] — Hazard ratio and CIs were computed from a stratified Cox model according to stratification factors as per IRT

5. Secondary Outcome: TTD in Physical Function as Determined by European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Cancer-specific Module With 30 Items (EORTC QLQ C30)
Description: TTD was defined as time from baseline(Cycle 1,Day 1) until first ≥10-point change from baseline up to end of treatment assessment before initiation of further anticancer therapy and analysis cut-off date.For TTD in physical function from EORTC QLQ-C30, deterioration=decrease of at least 10 points from baseline score.EORTC QLQ-C30(C30) is 30-item, cancer specific that includes global health status/health-related quality of life(GHS/QoL), functional scales(physical,role,emotional,cognitive,social), symptom scales(fatigue,nausea&vomiting,pain), 5 symptom items(dyspnea,insomnia,appetite loss,constipation,diarrhea,perceived financial difficulties). Most questions from QLQ-C30 were rated on 4-point scale(1/Not at All to 4/Very Much), except Items 29-30,which comprise GHS scale and were rated on 7-point scale(1/Very Poor to 7/Excellent). All scales were transformed from raw scores to linear scales ranging 0-100. High score represented favorable outcome with best quality of life.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tusamitamab Ravtansine | Docetaxel
Number analyzed (Participants) | 194 | 195
months | 7.46 [5.552 to 15.211] | 4.17 [3.023 to 4.567]
Statistical Analysis 1: Comparison: Tusamitamab Ravtansine vs Docetaxel; Test type: Superiority; p = 0.0002, Log Rank — P-value is provided for information only, there is no statistical inference based on this P-value; Hazard Ratio (HR) = 0.544, 95% CI 2-sided [0.388 to 0.763] — Hazard ratio and CIs were computed from a stratified Cox model according to stratification factors as per IRT

6. Secondary Outcome: TTD in Role Function Measured by EORTC QLQ C30
Description: TTD was defined as time from baseline (Cycle 1, Day 1) until first ≥10-point change from baseline up to end of treatment assessment before initiation of further anticancer therapy and analysis cut-off date. For TTD in role function from EORTC QLQ-C30, deterioration = decrease of at least 10 points from baseline score. EORTC QLQ-C30 (C30) is a 30-item, cancer specific that includes GHS/QoL, functional scales (physical, role, emotional, cognitive, social), symptom scales (fatigue, nausea & vomiting, pain), 5 symptom items (dyspnea, insomnia, appetite loss, constipation, diarrhea, perceived financial difficulties item). Most questions from QLQ-C30 were rated on a 4-point scale (1/Not at All to 4/Very Much), except Items 29-30, which comprise GHS scale and were rated on a 7-point scale (1/Very Poor to 7/Excellent). All scales were transformed from raw scores to linear scales ranging 0 to 100. A high score represented a favorable outcome with a best quality of life for participant.
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tusamitamab Ravtansine | Docetaxel
Number analyzed (Participants) | 194 | 195
months | 5.55 [3.713 to 6.308] | 4.17 [2.793 to 4.370]
Statistical Analysis 1: Comparison: Tusamitamab Ravtansine vs Docetaxel; Test type: Superiority; p = 0.0305, Log Rank — P-value is provided for information only, there is no statistical inference based on this P-value; Hazard Ratio (HR) = 0.735, 95% CI 2-sided [0.533 to 1.014] — Hazard ratio and CIs were computed from a stratified Cox model according to stratification factors as per IRT

7. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A SAE was defined as any untoward medical occurrence that, at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event. TEAEs were defined as AEs that developed, worsened, or became serious during the treatment period.
Time Frame: From date of first study treatment administration (Day 1) up to 30 days after the last dose of study treatment administration, up to 151 weeks
Reporting Status: Not Posted, anticipated posting 2027-08

8. Secondary Outcome: Number of Participants With Potentially Clinically Significant Abnormalities (PCSA) in Hematology Parameters
Description: Blood samples were collected to determine the abnormalities in hematology parameters.
Time Frame: as for outcome 7
Reporting Status: Not Posted, anticipated posting 2027-08

9. Secondary Outcome: Number of Participants With PCSA in Clinical Chemistry
Description: Blood samples were collected to determine the clinical chemistry laboratory abnormalities.
Time Frame: as for outcome 7
Reporting Status: Not Posted, anticipated posting 2027-08

10. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the date of first initial occurrence of a CR or PR to the date of first documentation of objective PD according to RECIST 1.1 before the initiation of any posttreatment anticancer therapy or death due to any cause, whichever occurred first. CR was defined as disappearance of all target and non-target lesions, and normalization of tumor marker level. Any pathological lymph nodes (whether target or non-target) must have had reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. PD was defined as unequivocal progression of existing non-target lesions; appearance of 1 or more new lesions; at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Tumor assessments performed at screening, and every 8 weeks +/-5 days thereafter, up to 189 weeks
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tusamitamab Ravtansine | Docetaxel
Number analyzed (Participants) | 41 | 45
months | 11.07 [5.158 to 19.844] | 5.75 [4.074 to 7.326]

ADVERSE EVENTS:
Time Frame: TEAEs were collected from date of first study treatment administration (Day 1) up to 30 days after the last dose of study treatment administration, up to 151 weeks. All-cause mortality data was collected from date of first study treatment administration (Day 1) until the primary analysis date of 22 September 2023 (up to 189 weeks).
Description: Analysis was performed on safety population. All-cause mortality data was collected on randomized population.
Arm/Group | Tusamitamab Ravtansine | Docetaxel
All-Cause Mortality (participants affected / at risk) | 109/194 | 110/195
Serious Adverse Events (participants affected / at risk) | 55/194 | 68/177
Other Adverse Events (participants affected / at risk) | 159/194 | 151/177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tusamitamab Ravtansine (N=194) | Docetaxel (N=177)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 11 (11)
Myelosuppression (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 4 (5)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo Positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Dry Eye (Eye disorders) | 1 (1) | 0 (0)
Uveitis (Eye disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 4 (4)
Colitis Ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis Ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastric Ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal Inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 2 (2)
Mechanical Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Obstruction Gastric (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal Stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Disease Progression (General disorders) | 7 (7) | 3 (3)
Fatigue (General disorders) | 0 (0) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Sudden Death (General disorders) | 1 (1) | 2 (2)
Cholecystitis Acute (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic Failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abdominal Abscess (Infections and infestations) | 0 (0) | 1 (1)
Abdominal Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Atypical Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 2 (2) | 2 (2)
Covid-19 Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Clostridium Difficile Infection (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal Infection (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Infectious Pleural Effusion (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Neutropenic Infection (Infections and infestations) | 0 (0) | 3 (3)
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 8 (8)
Pneumonia Influenzal (Infections and infestations) | 1 (1) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Accidental Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Compression Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 0 (0)
Blood Creatinine Increased (Investigations) | 0 (0) | 1 (1)
Neutrophil Count Decreased (Investigations) | 0 (0) | 2 (2)
Oxygen Saturation Decreased (Investigations) | 0 (0) | 1 (1)
Platelet Count Decreased (Investigations) | 1 (1) | 0 (0)
Transaminases Increased (Investigations) | 0 (0) | 1 (1)
Troponin T Increased (Investigations) | 1 (1) | 0 (0)
White Blood Cell Count Decreased (Investigations) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Spinal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intracranial Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant Pleural Effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pericardial Effusion Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour Associated Fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain Oedema (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Generalised Tonic-Clonic Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial Pressure Increased (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Malignant Spinal Cord Compression (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax Spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Peripheral Artery Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tusamitamab Ravtansine (N=194) | Docetaxel (N=177)
Neutropenia (Blood and lymphatic system disorders) | 3 (4) | 10 (12)
Decreased Appetite (Metabolism and nutrition disorders) | 39 (40) | 41 (51)
Insomnia (Psychiatric disorders) | 8 (9) | 14 (14)
Dysgeusia (Nervous system disorders) | 5 (6) | 15 (17)
Headache (Nervous system disorders) | 8 (8) | 9 (10)
Neuropathy Peripheral (Nervous system disorders) | 11 (11) | 7 (14)
Paraesthesia (Nervous system disorders) | 17 (18) | 6 (7)
Peripheral Sensory Neuropathy (Nervous system disorders) | 15 (18) | 15 (15)
Cataract (Eye disorders) | 11 (12) | 3 (3)
Dry Eye (Eye disorders) | 11 (12) | 7 (7)
Keratitis (Eye disorders) | 21 (27) | 1 (1)
Keratopathy (Eye disorders) | 31 (38) | 2 (2)
Lacrimation Increased (Eye disorders) | 2 (2) | 10 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 17 (19)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 (18) | 18 (21)
Abdominal Pain (Gastrointestinal disorders) | 12 (14) | 7 (7)
Constipation (Gastrointestinal disorders) | 21 (21) | 21 (27)
Diarrhoea (Gastrointestinal disorders) | 29 (34) | 49 (58)
Nausea (Gastrointestinal disorders) | 26 (35) | 37 (44)
Stomatitis (Gastrointestinal disorders) | 6 (6) | 22 (27)
Vomiting (Gastrointestinal disorders) | 10 (13) | 19 (22)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 59 (60)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (15) | 9 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 (24) | 16 (19)
Back Pain (Musculoskeletal and connective tissue disorders) | 19 (19) | 13 (15)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (11) | 11 (17)
Asthenia (General disorders) | 32 (38) | 41 (54)
Fatigue (General disorders) | 26 (52) | 37 (44)
Oedema Peripheral (General disorders) | 7 (8) | 34 (35)
Pyrexia (General disorders) | 12 (14) | 17 (20)
Neutrophil Count Decreased (Investigations) | 1 (4) | 10 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2023-03-13): https://cdn.clinicaltrials.gov/large-docs/56/NCT04154956/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-28): https://cdn.clinicaltrials.gov/large-docs/56/NCT04154956/SAP_001.pdf